CLINICAL TRIAL: NCT02515539
Title: Early Feasibility Study of the CardiAQ™ Transcatheter Mitral Valve Implantation (TMVI) System (Transfemoral and Transapical Delivery Systems)
Brief Title: Early Feasibility Study of the CardiAQ™ TMVI System (Transfemoral and Transapical DS)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Edwards Lifesciences terminated the IDE associated with this study. No patients enrolled.
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-3103-01
Record Dates: First submitted 2015-08-03; First posted 2015-08-04 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2015-08

CONDITIONS: Mitral Insufficiency; Heart Valve Disease; Cardiovascular Disease; Heart Disease
Keywords: Transcatheter Mitral Valve Replacement; Mitral Regurgitation; Mitral Insufficiency; Transapical; Transfemoral
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CardiAQ TMVI System (Transapical & Transfemoral DS) (Experimental): CardiAQ TMVI System using either the Transapical or Transfemoral Delivery System
  Interventions: Device: CardiAQ TMVI System (Transapical & Transfemoral DS)

INTERVENTIONS:
Device: CardiAQ TMVI System (Transapical & Transfemoral DS) — CardiAQ TMVI System using either the Transapical or Transfemoral Delivery System

SUMMARY:
The purpose of the study is to generate early US feasibility data of the CardiAQ™ Transcatheter Mitral Valve Implant System.

The study will enroll patients with moderate to severe mitral valve regurgitation who are considered high risk for mortality and morbidity from conventional open-heart surgery.

DETAILED DESCRIPTION:
Early feasibility study - multi-center, prospective, single-arm, and non-randomized study without concurrent or historical controls.

The primary objective of the study is to generate early feasibility data for the CardiAQ™ Transcatheter Mitral Valve Implant System with the Transfemoral and Transapical Delivery Systems for the treatment of moderate to severe mitral valve regurgitation in patients who are considered high risk for mortality and morbidity from conventional open-heart surgery.

The secondary objectives of the study are to evaluate the long-term safety of the device and the effects of the device on performance, functional, quality of life parameters, and technical, device, procedural, and individual patient successes.

The study is to be performed at a maximum of 5 investigational sites in the US.

ELIGIBILITY:
Key Inclusion Criteria:

* NYHA Classification ≥ III
* Left Ventricular Ejection Fraction ≥ 30%
* Mitral Regurgitation ≥ Grade 3+
* Subject meets anatomical and eligibility criteria for the investigational device

Exclusion Criteria:

* See Protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Composite Major Adverse Event Rate | 30-Day

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Szeto, MD, Principal Investigator — University of Pennsylvania; Howard Herrmann, MD, Principal Investigator — University of Pennsylvania; Saibal Kar, MD, Principal Investigator — Cedars-Sinai Medical Center; Alfredo Trento, MD, Principal Investigator — Cedars-Sinai Medical Center